CLINICAL TRIAL: NCT01397656
Title: Comparison of Bystander Fatigue and CPR Quality When Using the 2010 Continuous Chest Compression Versus the 2005 30:2 Chest Compression to Ventilation Resuscitation Guidelines for Laymen: A Randomized Crossover Trial
Brief Title: Bystander Fatigue and CPR Quality Using Continuous Compressions Versus 30:2 Compressions to Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2011358-01H
Record Dates: First submitted 2011-06-13; First posted 2011-07-19 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2017-06

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; CPR; resuscitation; fatigue; quality
MeSH Terms: conditions — Heart Arrest; Fatigue | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPR 30:2 (Active Comparator): 30 chest compressions to 2 ventilations followed by cross-over to CPR with Continuous Compressions
  Interventions: Procedure: CPR using 30:2 ratio
- CPR with Continuous Compressions (Active Comparator): Continuous Chest Compressions without ventilation followed by CPR 30:2 (30 chest compressions to 2 ventilations)
  Interventions: Procedure: CPR using continuous compressions

INTERVENTIONS:
Procedure: CPR using 30:2 ratio — Participants will begin performing CPR using a ratio of 30 compressions to 2 ventilations. Participants will then cross over to the other intervention and use continuous compressions.
  Other Names: cardiopulmonary resuscitation
  Arms: CPR 30:2
Procedure: CPR using continuous compressions — Participants will begin performing CPR using continuous chest compressions. Participants will then cross-over to the other intervention arm and perform CPR using a ratio of 30 compressions to 2 ventilations.
  Other Names: cardiopulmonary resuscitation
  Arms: CPR with Continuous Compressions

SUMMARY:
STUDY OBJECTIVES The overall goal of this study is to compare bystander fatigue and CPR quality after 5 minutes of continuous chest compressions versus the 2005 30:2 chest compression to ventilation Resuscitation Guidelines, in a population aged 55 or greater.

More specifically, the investigators will compare each CPR ratio with regard to:

1. The achieved frequency and depth of chest compressions, and
2. Participant rating of their perceived level of exertion.

STUDY HYPOTHESIS

In a population aged 55 or greater, the new CPR recommendations will lead to:

1. less frequent and shallower chest compressions over the 5-minute study period; and
2. higher rating of perceived level of exertion when compared to the 2005 30:2 CPR ratio.

DETAILED DESCRIPTION:
Background: Cardiac arrest is the number one cause of mortality in the Canadian population. Out-of-hospital bystander cardiopulmonary resuscitation (CPR) is associated with a 3 to 4 fold increase in survival for cardiac arrest, but citizens are often reluctant to initiate CPR because of its mouth-to-mouth component. In an effort to increase bystander CPR rates in the community and minimize interruptions in chest compressions, the 2010 Resuscitation Guidelines changed the 2005 recommended 30:2 compression to ventilation ratio to continuous chest compressions for laymen. Although the 30:2 ratio is meant to increase survival for cardiac arrest, the ability of rescuers to deliver continuous chest compressions has never been studied. Little is known about the impact of the new recommendations on bystander fatigue and resulting CPR quality.

Objectives: The overall goal of this study is to compare bystander fatigue and CPR quality after 5 minutes continuous chest compressions versus the 2005 30:2 chest compression to ventilation Resuscitation Guidelines in a population aged 55 or greater.

More specifically, the investigators will compare each CPR ratio with regard to:

1. The achieved frequency and depth of chest compressions, and
2. Participants' rating of their perceived level of exertion.

Methods: The investigators will conduct a randomized cross-over trial comparing bystander fatigue and CPR quality using two different CPR ratios. Intervention: All participants will be asked to perform two 5-minute sessions of CPR on a manikin - one session using the 30:2 ratio, the other using continuous chest compressions. There will be a supervised practice session in the beginning, and resting periods in between. The order in which the sessions will be executed will be determined in a random fashion. The study population will consist of volunteers aged 55 or older, a group most susceptible to perform CPR on a real victim. The study will take place in a busy public area of The Ottawa Hospital, Civic Campus, and in senior's activity centres in Ottawa. Participants will have to score 3 or less on the validated Clinical Frailty Scale in order to participate in the study. Participants with physical limitations or disease processes precluding their ability to safely perform CPR will be excluded. Outcome measures: Information on age, gender, prior CPR training, and measure of frailty will be collected at the time of enrollment. The number, frequency, and quality of chest compressions (depth and release) will be measured during each CPR session using a Zoll cardiac monitor with the ability to measure CPR processes. Heart rate and blood pressure will be measured before and after each CPR session. The participants will be asked to rate their level of fatigue before and after each CPR session using the validated Borg Rating of Perceived Exertion scale. Sample size: The investigators hope to recruit 60 participants. Data analysis for Objective#1 will include descriptive statistics and a paired t-test with 95% confidence interval; Objective#2 will be analyzed using descriptive statistics and Wilcoxon Rank Sum test. In addition, as an exploratory analysis, the investigators also assessed the rate of change over time in the number of chest compressions performed adequately using a random coefficient model. This study protocol will be reviewed by the OHREB before implementation, and will be entered in a trial registry.

Importance of the study: Data from this study will evaluate bystander fatigue and resulting CPR quality when comparing the 2010 continuous chest compression to the 2005 30:2 chest compression to ventilation Resuscitation Guidelines. This project will improve our understanding of the physiological demands associated with the implementation of the new CPR Resuscitation Guidelines for laymen. The investigators anticipated the results from this study will be widely distributed, and will help shape the 2015 iteration of the Resuscitation Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female person aged 55 or older
* Must score 3 or less on the validated Clinical Frailty Scale
* Able to follow instructions in English or French
* Able to understand and give informed consent

Exclusion Criteria:

* Musculoskeletal condition precluding the ability to kneel down and perform CPR (e.g. severe arthritis, cast, wrist sprain, recent joint surgery)
* Cardiovascular condition precluding the ability to perform a moderate effort (e.g. myocardial infarction or cardiovascular procedure in the last 3 months, recurrent angina, chest pain under investigation)
* Pulmonary condition precluding the ability to perform a moderate effort (e.g. emphysema, severe asthma, pneumonia)
* Active communicable disease (e.g. tuberculosis, meningitis, gastro enteritis, hepatitis A or B, herpes simplex)
* Inability to perform chest compressions at appropriate rate and depth despite positive feedback during one to two-minute practice session

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Civic Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vaillancourt C, Midzic I, Taljaard M, Chisamore B. Performer fatigue and CPR quality comparing 30:2 to 15:2 compression to ventilation ratios in older bystanders: A randomized crossover trial. Resuscitation. 2011 Jan;82(1):51-6. doi: 10.1016/j.resuscitation.2010.09.003. Epub 2010 Oct 14. PMID 20947241
- [Result] Liu S, Vaillancourt C, Kasaboski A, Taljaard M. Bystander fatigue and CPR quality by older bystanders: a randomized crossover trial comparing continuous chest compressions and 30:2 compressions to ventilations. CJEM. 2016 Nov;18(6):461-468. doi: 10.1017/cem.2016.373. Epub 2016 Sep 21. PMID 27650514

RESULTS

PARTICIPANT FLOW:
Groups:
- CPR 30:2 Then CPR With Continuous Compressions: 30 chest compressions to 2 ventilations, then continuous chest compressions
  Bystander CPR using 30:2 ratio versus continuous compression: Participants will use 2 CPR techniques, one with 30 compressions to 2 ventilations and the other with continuous compressions without ventilation
- CPR With Continuous Compressions Then CPR 30:2: Continuous Chest Compressions without ventilation then CPR using 30:2 ratio
  Bystander CPR using 30:2 ratio versus continuous compression: Participants will use 2 CPR techniques, one with 30 compressions to 2 ventilations and the other with continuous compressions without ventilation
Period: Overall Study
Arm/Group | CPR 30:2 Then CPR With Continuous Compressions | CPR With Continuous Compressions Then CPR 30:2
Started | 33 | 30
Completed | 33 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CPR 30:2 Then CPR With Continuous Compressions: 30 chest compressions to 2 ventilations
  Bystander CPR using 30:2 ratio versus continuous compression: Participants will use 2 CPR techniques, one with 30 compressions to 2 ventilations and the other with continuous compressions without ventilation
- CPR With Continuous Compressions Then CPR 30:2: Continuous Chest Compressions without ventilation
  Bystander CPR using 30:2 ratio versus continuous compression: Participants will use 2 CPR techniques, one with 30 compressions to 2 ventilations and the other with continuous compressions without ventilation
- Total: Total of all reporting groups
Arm/Group | CPR 30:2 Then CPR With Continuous Compressions | CPR With Continuous Compressions Then CPR 30:2 | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (6.5) | 69.9 (6.3) | 70.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 30 | 63
CPR Training [Count of Participants; unit: Participants] | 18 | 20 | 38
CPR Experience [Count of Participants; unit: Participants] — Prior experience delivering CPR
  Participants | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: CPR Quality
Description: Count of compressions at a depth over 2 inches
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: Compressions
Groups:
- CPR 30:2: 30 chest compressions to 2 ventilations
- CPR With Continuous Compressions: Continuous Chest Compressions without ventilation
  Bystander CPR using 30:2 ratio versus continuous compression: Participants will use 2 CPR techniques, one with 30 compressions to 2 ventilations and the other with continuous compressions without ventilation
Arm/Group | CPR 30:2 | CPR With Continuous Compressions
Number analyzed (Participants) | 62 | 63
Compressions | 324.9 (120) | 381.5 (68.5)

2. Secondary Outcome: Heart Rate
Time Frame: Assessed immediately before and after 5 minutes of CPR
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- CPR With Continuous Compressions: Continuous Chest Compressions without ventilation
Arm/Group | CPR 30:2 | CPR With Continuous Compressions
Number analyzed (Participants) | 62 | 63
beats per minute | 82.8 (16.1) | 82.4 (15.1)

3. Secondary Outcome: Blood Pressure
Description: Mean arterial pressure (mmHg)
Time Frame: Assessed immediately before and after 5 minutes of CPR
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CPR 30:2 | CPR With Continuous Compressions
Number analyzed (Participants) | 62 | 63
mmHg | 109.8 (10.7) | 110.3 (11.5)

4. Secondary Outcome: Borg Rating of Perceived Exertion Scale
Description: The Borg Rating of Perceived Exertion scale ranges from 6-20, where a score of 6 is associated with the least fatigue
Time Frame: Assessed immediately before and after 5 minutes of CPR
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CPR With Continuous Compressions: Continuous Chest Compressions
Arm/Group | CPR 30:2 | CPR With Continuous Compressions
Number analyzed (Participants) | 62 | 63
units on a scale | 11.0 (2.6) | 11.6 (3.0)

ADVERSE EVENTS:
Arm/Group | CPR 30:2 Then CPR With Continuous Compressions | CPR With Continuous Compressions Then CPR 30:2
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No